CLINICAL TRIAL: NCT00162435
Title: Warfarin Induction Regimen Based Upon CYP2C9, VKORC1 Factor VII Genotyping, PMR and INR Monitoring, as Compared to the Conventional Regimen: a Prospective Controlled Study
Brief Title: Genetic Determinants of Warfarin Anticoagulation Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: United States - Israel Binational Science Foundation (Other); Israel Science Foundation (Other); Ministry of Health, Israel (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: yc19553-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-03

CONDITIONS: Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation | interventions — Warfarin

ARMS (2):
- Genetic (Experimental)
  Interventions: Drug: Warfarin
- Control (Experimental)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin

SUMMARY:
The response to warfarin varies greatly among individuals. Some of this variability can be ascribed to genetic polymorphisms in the gene encoding for CYP2C9, the enzyme mediating the metabolism of S warfarin. In addition genetic polymorphism in other genes (i.e. VKORC1, factor VII) have been shown to account for some of the variability in the response to warfarin irrespective of CYP2C9.The present study has several segments:

1. Evaluation of the relationship between genetic polymorphisms in the genes encoding for CYP2C9, VKORC1 and factor VII and warfarin maintenance dose at steady state. This study is a confirmation of previous data in our own population.
2. Evaluation of relationship between genetic polymorphisms in the genes encoding for CYP2C9, VKORC1 and factor VII and warfarin loading dose during the induction period.
3. Testing the hypothesis that warfarin loading based on the individual's combined CYP2C9, VKORC1 and factor VII genotype may be more efficient and associated with reduced adverse drug effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom warfarin is about to be initiated
* Desired therapeutic range >2 and <3

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2002-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic end points: | 1-4 months
Warfarin clearance and formation clearance of 7-hydroxy-warfarin at steady state | 1-4 months
Pharmacodynamic. | 1-4 months
Maintenance dose of warfarin at steady state. | 1-4 months
Time to reach INR > 2. | 1-4 months
Time to reach pharmacodynamic steady state. | 1-4 months
Time spent at therapeutic INR <3 and >2. | 1-4 months
Time spent at INR >3. | 1-4 months
Time spent at INR <2. | 1-4 months
The incidence of minor and major bleeding episodes. | 1-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Caraco Y, Blotnick S, Muszkat M. CYP2C9 genotype-guided warfarin prescribing enhances the efficacy and safety of anticoagulation: a prospective randomized controlled study. Clin Pharmacol Ther. 2008 Mar;83(3):460-70. doi: 10.1038/sj.clpt.6100316. Epub 2007 Sep 12. PMID 17851566